CLINICAL TRIAL: NCT03967366
Title: Association Between Plasma Melatonin and Coronary Artery Calcification
Brief Title: Melatonin and Coronary Artery Calcification
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Chen Wei Ren, MD, Prof., Chinese PLA General Hospital
Other Study IDs: MelandCAC
Record Dates: First submitted 2019-05-26; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Calcification
Keywords: Melatonin; coronary artery calcification; relation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood samples were acquired to evaluate the melatonin, high sensitivity C-reactive protein, malondialdehyde level.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- plasma melatonin 1: Quartile 1 of plasma melatonin
- plasma melatonin 2: Quartile 2 of plasma melatonin
- plasma melatonin 3: Quartile 3 of plasma melatonin
- plasma melatonin 4: Quartile 4 of plasma melatonin

SUMMARY:
The investigators planned to research the association between plasma melatonin and coronary artery calcification in a Chinese population.

DETAILED DESCRIPTION:
Coronary artery calcification (CAC) is prevalent in coronary artery disease (CHD), and the extent of CAC predicts cardiovascular risk. The causes of CAC include dysregulated matrix metabolism, epitaxial mineral deposition, inflammation, oxidative stress, and apoptosis. Melatonin is the main indoleamine produced by the pineal gland; it is known recently to have anti-inflammatory, anti-cancer and antioxidant activities. Several studies have shown that melatonin protects against inflammation and apoptosis in vascular calcification. Melatonin also inhibits oxidative stress-induced apoptosis and calcification in endplate chondrocytes. However, no study has evaluated whether melatonin is associated with CAC in patients with coronary atherosclerosis. The investigators planned to research the association between plasma melatonin and coronary artery calcification.

ELIGIBILITY:
Inclusion Criteria:

Patients with angina-like chest pain, were included in this study. All subjects had blood samples collected and all underwent a coronary CTA scan.

Exclusion Criteria:

1. melatonin treatment
2. coronary revascularization (percutaneous coronary intervention or coronary artery bypass graft surgery)
3. heart failure or cardiomyopathies
4. hepatic failure
5. renal dysfunction
6. haemolytic disorders
7. thyroid disease
8. neoplastic diseases
9. acute infectious or inflammatory conditions.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: PLA general hospital (PLAGH) is a large national tertiary-care center in the Beijing, China. The investigators enrolled patients consecutively in PLAGH.
Sampling Method: Probability Sample
Enrollment: 574 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
correlations of CAC score with melatonin concentrations | Subjects underwent a CAC scan at baseline.
  CAC score was obtained using the coronary CTA and Agatston score.

SECONDARY OUTCOMES:
correlations of CAC score with high-sensitivity C-reactive protein (hsCRP) level | Subjects had blood samples collected at baseline.
  The hsCRP levels were analyzed by a sandwich enzyme linked immunosorbent assay.
correlations of CAC score with malondialdehyde (MDA) level | Subjects had blood samples collected at baseline.
  The MDA levels were analyzed by a sandwich enzyme linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Overall Officials: yu jie zhou, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- PLA general hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olson F, Engborg J, Gronhoj MH, Sand NP, Lambrechtsen J, Steffensen FH, Nybo M, Gerke O, Mickley H, Diederichsen AC. Association between high-sensitive troponin I and coronary artery calcification in a Danish general population. Atherosclerosis. 2016 Feb;245:88-93. doi: 10.1016/j.atherosclerosis.2015.12.017. Epub 2015 Dec 15. PMID 26714045
- [Background] Kim HJ, Kim JH, Joo MC. Association of Exercise Capacity, Cardiac Function, and Coronary Artery Calcification with Components for Metabolic Syndrome. Biomed Res Int. 2018 Oct 4;2018:4619867. doi: 10.1155/2018/4619867. eCollection 2018. PMID 30402479
- [Background] Zhao X, Zhang HW, Li S, Zhang Y, Xu RX, Zhu CG, Wu NQ, Guo YL, Qing P, Li XL, Liu G, Dong Q, Sun J, Li JJ. Association between plasma proprotein convertase subtisilin/kexin type 9 concentration and coronary artery calcification. Ann Clin Biochem. 2018 Jan;55(1):158-164. doi: 10.1177/0004563217695351. Epub 2017 May 15. PMID 28166668
- [Background] Fernandez A, Ordonez R, Reiter RJ, Gonzalez-Gallego J, Mauriz JL. Melatonin and endoplasmic reticulum stress: relation to autophagy and apoptosis. J Pineal Res. 2015 Oct;59(3):292-307. doi: 10.1111/jpi.12264. Epub 2015 Aug 9. PMID 26201382